CLINICAL TRIAL: NCT00108212
Title: Clinical Implications of Genetic Alterations in TG Rich Lipoproteins
Brief Title: Effect of Diet on Men and Women With Genetic Alterations Associated With Abnormal Blood Tests
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CARD-005-03S
Record Dates: First submitted 2005-04-14; First posted 2005-04-15 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2007-04

CONDITIONS: Dyslipidemia
Keywords: Diet; triglyceride; inflammation; Genetic polymorphism
MeSH Terms: conditions — Dyslipidemias; Inflammation | interventions — Diet

INTERVENTIONS:
Behavioral: Diet

SUMMARY:
The purpose of this study is to evaluate different diets and the effects of blood measures or inflammation and endothelial function in association with genetics tending to abnormal blood test levels.

ELIGIBILITY:
Inclusion Criteria:

* Polymorphism in Apo C3 promoter and normal controls.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 2005-01; Study Completion 2007-12

CONTACTS AND LOCATIONS:
Locations (1):
- VA Maryland Health Care System, Baltimore, Maryland, United States